CLINICAL TRIAL: NCT03873454
Title: The Effects of Music on Perioperative Outcomes in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Anaesthesia, Principal Investigator, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIRB 2014/378/D
Record Dates: First submitted 2014-08-12; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cataract Surgery; Stress Levels; Music Improving Outcomes in Cataract Surgery
Keywords: cataract surgery; music; salivary cortisol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental Group (Active Comparator): The experimental group listened to music and wore Sennheiser non-occlusive headphones
  Interventions: Device: Sennheiser non-occlusive headphones
- Control 1 with no music (Other): This cohort wore non-occlusive earphones but did not listen to music
  Interventions: Device: Sennheiser non-occlusive headphones without music
- Control 2 with no music (Other): The control 2 patients did not listen to music nor wore earphones.
  Interventions: Other: No Sennheiser non-occlusive headphones

INTERVENTIONS:
Device: Sennheiser non-occlusive headphones — Patients listened to music of their choice using non-occlusive headphones
  Arms: Experimental Group
Device: Sennheiser non-occlusive headphones without music — Patients wore non-occlusive headphones but had no music playing
  Arms: Control 1 with no music
Other: No Sennheiser non-occlusive headphones — Patients did not wear non-occlusive headphones and did not listen to music
  Arms: Control 2 with no music

SUMMARY:
The hypothesis of this trial is that listening to music will decrease the stress levels that patients face as evidenced by their STAI scores, salivary cortisol levels and intra-operative autonomic parameters.

DETAILED DESCRIPTION:
This randomized control trial was conducted from May- July 2014 across National University Hospital and Singapore National Eye Centre. All the patients of 10 consultants and senior consults and X medical officers were included in the study. A total of 148 participants were surveyed, and a total of X saliva samples were collected.

The inclusion criterion for patients was cataract surgery patients aged 50 years and above, with an acceptable hearing level based on CALFRAST hearing and the ability to wear clip-on on-ear headphones without discomfort. They were required to be mentally and physically capable of informed consent. Patients were also required to be ASA Grade 3 or lower.

Inclusion criterion for surgeons was surgeons doing phacoemulsification cataract surgeries, and for anaesthetists, the inclusion criteria was anaesthetists using only minimal sedation for the procedure.

Exclusion criteria was severe/profound hearing impairments, patients with intellectual disabilities, patients on psychotropic medications or drugs affecting mood or hemodynamic status, ASA grade 4 and parturients

Exclusion criterion for surgeons included ECCE procedures. Exclusion criteria for anaesthetists was anaesthetists using moderate sedation, or who used non-standard drugs including Droperidol.

Both the NHG Domain-Specific Institutional Review Board and the Singhealth Institutional Review Board approved the study in May 2014, and all ethical consideration complied with. Written informed consent was sought prior to the questionnaire administration, and participants were allowed to withdraw from the study at any time during data collection.

The study had 3 arms- an experimental group of patients who listened to music via headphones, a first control group of patients who wore earphones but did not listen to music, and a second control group of patients who neither listened to music nor wore headphones. All patients were assigned a study number and no patient identifiers were noted.

1 hour before the procedure, study participants were approached to do an anonymous survey. Patients were then asked to produce a saliva sample by pooling saliva under the tongue for 5 minutes.

Finally, patients in the experimental group choose one of 30 playlists; if a patient did not find a playlist to their satisfaction, Spotifiy® was used to generate a new playlist. Patients were also allowed to listen to their preferred local radio station. Music was played using wireless headphones synced with a Jabra® Bluetooth device which was clipped onto the patients OT gown.

Intra-operatively, both the surgeon and anaesthetist were blinded to what arm of the study the patient was undergoing. Autonomic parameters (blood pressure, Mean Arterial Pressure, Respiratory Rate and Heart Rate) as well as dosages of drugs administered (anxiolytics, sedatives, anaesthetics, any other drugs used). The total time for the procedure was noted. Post-operatively, the surgeon was surveyed for complexity of the case and ease of communication with the patient, whilst the anaesthetist was surveyed for depth of anaesthesia and ease of communication with the patient.

10 minutes post-procedurally, the patient was surveyed again and saliva samples were collected.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery patients aged 50 years and above, with an acceptable hearing level based on CALFRAST hearing and the ability to wear clip-on on-ear headphones without discomfort. They were required to be mentally and physically capable of informed consent. Patients were also required to be ASA Grade 3 or lower.
* Surgeons doing phacoemulsification cataract surgeries, and for anaesthetists, the inclusion criteria was anaesthetists using only minimal sedation for the procedure.

Exclusion Criteria:

* Severe/profound hearing impairments, patients with intellectual disabilities, patients on psychotropic medications or drugs affecting mood or hemodynamic status, ASA grade 4 and parturients
* Exclusion criterion for surgeons included ECCE procedures. Exclusion criteria for anaesthetists was anaesthetists using moderate sedation, or who used non-standard drugs including Droperidol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol | Pre-operatively
  1 hour before the surgery a saliva sample was collected from the patient in order to test for salivary cortisol as a measure of stress.
Salivary Cortisol | 10 minutes post-operatively
  10 minutes after the surgery, a saliva sample was collected from the patient in order to test for salivary cortisol as a measure of stress.

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof Lian Kah Ti, MBBS, MMED, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore National Eye Centre, Singapore